CLINICAL TRIAL: NCT05843357
Title: PAPSY: Snadné zjištění Poruch paměti pomocí Velmi krátkých testů ALBA a POBAV u psychiatrických diagnóz v celé ČR
Brief Title: PAPSY - Memory in Psychiatry
Acronym: PAPSY
Status: Active, not recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Tadeáš Mareš, Consultation-liaison psychiatrist, Charles University, Czech Republic
Other Study IDs: PAPSY
Record Dates: First submitted 2023-03-15; First posted 2023-05-06 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Cognitive Impairment
Keywords: Cognitive Impairment; Outpatient Psychiatric Service; Population Distribution
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observed group: No intervention will be administered on behalf of the project. The participants will be tested using ALBA and PICNIR (non-invasive) cognitive tests, and further sFAQ-CZ and GDS-CZ questionnaires will be administered. Questionnaires FAQ-CZ and MBI-C-CZ will be distributed to participants´ caretakers.

SUMMARY:
Memory in Psychiatry project (PAPSY) aims to map the distribution and severity of cognitive impairment in patients of outpatient psychiatric offices across the geographical area of the Czech Republic. 1000 patients in 90 psychiatric offices will undergo cognitive tests (ALBA and PICNIR) and psychometric scales (sFAQ-CZ and GDS-CZ) to asses their functional state and depressive symptoms. If applicable, caretakers will also be asked about the extent of the participant's autonomy and behavioral impairment (using oFAQ-CZ and MBI-C-CZ scales).

The trial's primary goal is to assess the distribution of cognitive impairment among diagnostic groups in psychiatric care according to the ICD-10. Additionally, the feasibility of ALBA and PICNIR methods to uncover previously undiagnosed cognitive impairments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Dispensarization of at least six months in an outpatient psychiatric office with an ICD-10 diagnosis
* Age>=45
* Permanent residency in the geographical area of the Czech Republic

Exclusion Criteria:

* Diagnosis of mental retardation (F70-F79) according to ICD-10
* Refusal to sign the informed consent and consent with GDPR
* Uncorrected visual impairment
* Uncorrected auditory impairment
* Inability to participate in the project

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population is intended to be comprised of persons (45yrs+) living in the geographical area of the Czech Republic undergoing a treatment at an outpatient psychiatric office for a diagnosis defined in ICD-10 (excluding mental retardation). The probability sample will be created by a random selection of persons undergoing their regular outpatient psychiatric checkups.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Baseline ALBA | Established on Day 0 as a single assessment.
  Amnesia Light and Brief Assessment (ALBA) test is an innovative method to assess cognitive functions quickly. The cognitive performance is scaled as an overall score between 0-12 (a lower value denotes a more severe cognitive impairment).
Baseline PICNIR | Established on Day 0 as a single assessment.
  Picture Naming and Immediate Recall test (PICNIR) is an innovative test method to assess cognitive functions quickly. The cognitive performance is scaled as an overall score between 0-20 (a lower value denotes a more severe cognitive impairment).
Statistical analysis of ALBA results, | The final statistical analysis will be performed through study completion, an average of 6 months.
  Statistical analysis of ALBA results compared to groups determined by ICD-10 diagnosis and demographical data.
Statistical analysis of PICNIR results. | The final statistical analysis will be performed through study completion, an average of 6 months.
  Statistical analysis of PICNIR results compared to groups determined by ICD-10 diagnosis and demographical data.

SECONDARY OUTCOMES:
Baseline MBI-C-CZ | Established as a baseline on Day 0.
  Mild Behavioral Impairment - Checklist - Czech version (MBI-C-CZ) is a standardized questionnaire to assess behavioral impairment in 34 items. Each item is scaled between 0-3 (a higher value denotes a higher severity) to reach the overall score between 0-102 (a higher value denotes a higher overall severity of behavioral impairments)
Baseline sFAQ-CZ | Established as a baseline on Day 0.
  Functional Activities Questionnaire - Czech version (FAQ-CZ) is a standardized questionnaire administered to assess a patient´s functional state regarding daily activities. Ten items of daily functioning are scaled between 0-3 (a higher value denotes a higher dependency) to reach the overall score between 0-30 (a higher value denotes a higher dependency). This version of the scale will be used for participants´ self-evaluation.
Baseline GDS-CZ | Established as a baseline on Day 0.
  The Geriatric Depression Scale - Czech version (GDS-CZ) is a standardized questionnaire administered to assess depressive symptoms, particularly in the elderly population. Fifteen items are scaled between 0-1 to reach the overall score between 0-15 (a higher value denotes a higher level of depressive symptoms).
Baseline oFAQ-CZ | Established as a baseline on Day 0.
  Functional Activities Questionnaire - Czech version (FAQ-CZ) is a standardized questionnaire administered to assess a patient´s functional state regarding daily activities. Ten items of daily functioning are scaled between 0-3 (a higher value denotes a higher dependency) to reach the overall score between 0-30 (a higher value denotes a higher dependency). This version of the scale will be used for caretakers´ evaluation of participants´ functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Aleš Bartoš, M.D., Ph.D., Principal Investigator — Charles University, Czech Republic; Tadeáš Mareš, M.D., Principal Investigator — Charles University, Czech Republic
Locations (1):
- Teaching Hospital Královské Vinohrady, Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD is to be shared upon request by a verified researcher. The study director´s discretion is reserved.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon the final publication of the outcomes, indefinitely.
Access Criteria: Being a verified researcher.